CLINICAL TRIAL: NCT00555165
Title: A Prospective Multicenter Clinical Study of the Implantable Miniature Telescope* in Patients With Central Vision Impairment Associated With AMD: IMT-UK Protocol (*IMT by Dr. Isaac Lipshitz)
Brief Title: A Study of an Implantable Miniature Telescope in Patients With With End-Stage AMD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VisionCare, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IMT-UK
Record Dates: First submitted 2007-11-05; First posted 2007-11-07 (Estimated); Last update posted 2012-11-14 (Estimated); Status verified 2012-11

CONDITIONS: End Stage Macular Degeneration
Keywords: Macular Degeneration; Visual Impairment; Quality of Life; Implantable Telescope
MeSH Terms: conditions — Macular Degeneration; Vision Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- I (Experimental)
  Interventions: Device: Telescope prosthesis

INTERVENTIONS:
Device: Telescope prosthesis — Monocular implantation of the telescope prosthesis after cataract extraction

SUMMARY:
Evaluation of pre and post-implantation management of patients with end-stage age-related macular degeneration (AMD) who have been implanted with the implantable telescope (IMT) under CE Mark indicated use. This study is designed to evaluate in particular the optimal parameters for patient selection for use of this device in routine clinical practice.

ELIGIBILITY:
Inclusion Criteria:

CE Mark approved indication of use which includes

* At least 55 years of age
* Bilateral visual impairment due to geographic atrophy or disciform scars
* Evidence of cataract

Exclusion Criteria:

* Active CNV (or 'wet' AMD)
* Prior cataract or refractive surgery in the study eye

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2007-11; Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
Best-Corrected Visual Acuity | 1 year

SECONDARY OUTCOMES:
Quality of Life | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Giuliana Silvestri, MD FRCP FRCS, Principal Investigator — Royal Hospitals, Belfast Health & Social Care Trust
Locations (4):
- United Kingdom (4):
  - Frimley Park Hospital NHS Trust, Frimley, Surrey
  - Royal Hospitals, Belfast Health & Social Care Trust, Belfast
  - Moorfields Eye Hospital NHS Trust, London
  - King's College Hospital NHS Trust, London